CLINICAL TRIAL: NCT02315820
Title: Induction of Labor Versus Expectant Management of Large for Gestational Age/Macrosomic Babies at Term. A Multi-center Randomized Trial
Brief Title: Induction of Labor Versus Expectant Management of Large for Gestational Age/Macrosomic Babies at Term. A Multi-center Trial
Acronym: IOLEMMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Yuri perlitz, Director-High Risk Unit & Maternitiy department, The Baruch Padeh Medical Center, Poriya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: POR-0085-14
Record Dates: First submitted 2014-12-07; First posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Macrosomia; Induction of Labor; Expectant Management; Shoulder Dystocia
Keywords: Macrosomia; Induction of labor; Expectant management; Shoulder dystocia
MeSH Terms: conditions — Shoulder Dystocia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Induction of Labor (IOL) (Experimental): Group I, Induction of Labor group (IOL). Women will be admitted for induction at 38-40+3 weeks when estimated fetal weight 3800-4500 gram.
  Interventions: Procedure: Induction of labor group (Group I)
- Expectant (No Intervention): Group II. Will be expectantly managed until 40+6 weeks, or an induction indication will appear.

INTERVENTIONS:
Procedure: Induction of labor group (Group I) — Women at 38-40+3 weeks with estimated fetal weight 3800-4500 will be offered ripening and IOL.
  Arms: Induction of Labor (IOL)

SUMMARY:
The equipoise whether to Induce pregnant women with suspected large for gestational babies or suspected macrosomia babies at term pregnancy is not solved yet. Only 2 relatively small studies were conducted to answer this clinically important question.

The investigators will conduct a randomized controlled, multi-center study large enough to confirm or refute our assumption that induction of labor at term reduces the shoulder dystocia prevalence significantly compared to expectant management.

DETAILED DESCRIPTION:
Background: Macrosomia at term is associated with increased maternal and neonatal morbidity, including a higher rate of shoulder dystocia and cesarean section (CS). Induction of labor (IOL) has been suggested as a means to prevent further fetal weight gain and therefore to reduce possible neonatal and maternal complications which are related to fetal weight.

Working hypothesis and aims: The aims of this study are: 1) to determine whether or not IOL improves maternal and neonatal outcome in large for gestational age babies, 2) to determine maternal satisfaction from the labor and delivery process in both study groups. Our working hypothesis is that IOL will reduce the shoulder dystocia and CS rate of LGA\macrosomic babies at term.

Methods: Patient from 38+0 - 40+3 gestational weeks estimated fetal weight 3800 - 4500 gr will prospectively and randomly allocated into two groups: IOL (group I) and expectant management (group II). Women with diabetes, a previous cesarean delivery, or other contraindications for vaginal delivery or candidates for IOL for other reasons will be excluded from the study. Outcome variables will include shoulder dystocia, brachial plexus injury, bone fractures, cephalhematoma, intraventricular hemorrhage, cesarean delivery and other neonatal and maternal variables.

Expected results: IOL will reduce the shoulder dystocia and CS rate of LGA\macrosomic babies at term.

Importance: This randomized, prospective multicenter study addresses a prevalent clinical question which does not have an accurate answer in the medical literature. Current guidelines rely on small numbered patients, and are over 15 years old studies.

Probable implications to Medicine: This study will establish the right management for LAG\macrosomic babies at term, IOL or expectant management for spontaneous labor.

ELIGIBILITY:
Inclusion Criteria:

* Singleton,
* live fetus,
* Vx presentation,
* EFW 3800-4500 grams,
* eligible for vaginal delivery,
* signed the informed consent.

Exclusion Criteria:

* Pr. CS,
* Diabetes,
* fetal major malformations,
* maternal/fetal illness or condition requiring IOL.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 474 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Rate of shoulder dystocia | 3 years

SECONDARY OUTCOMES:
Neonatal morbidity composite outcome and maternal morbidity composite outcome. | 3 years
  For each study group a neonatal and maternal composite outcome will be presented. The neonatal composite outcome will include: Fetal death (before the onset of labor, during delivery, unknown), Neonatal death, Birth weight (grams), Apgar score 1 min, Apgar score 5 min, Cord PH, Shoulder dystocia, Erb palsy, 3rd/4th-degree lacerations, Intubation, CPAP or high-flow nasal cannula (HFNC) for ventilation. Neonatal encephalopathy, Seizures, Sepsis, Pneumonia, Meconium aspiration syndrome, Birth fractures, IVH, Hyperbilirubinemia requiring phototherapy or exchange transfusion. Hypoglycemia (gl<40) requiring IV therapy. Admission to NICU, Neonatal hospital stay. The maternal morbidity composite outcome will include: Chorioamnionitis PPH Maternal febrile morbidity requiring antibiotics administration. Anemia requiring blood transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Perlitz, MD, Principal Investigator — Director-High risk unit and maternal department

REFERENCES:
- [Derived] Boulvain M, Thornton JG. Induction of labour at or near term for suspected fetal macrosomia. Cochrane Database Syst Rev. 2023 Mar 8;3(3):CD000938. doi: 10.1002/14651858.CD000938.pub3. PMID 36884238